CLINICAL TRIAL: NCT04701385
Title: Plaque Erosion Prospective Study ii
Acronym: PEPSii
Status: Completed | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 270706
Record Dates: First submitted 2020-10-06; First posted 2021-01-08 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Atheroma; Myocardial
Keywords: Plaque Erosion; Circulating endothelial cells; Myocardial infarction; Neutrophils
MeSH Terms: conditions — Plaque, Atherosclerotic; Myocardial Infarction | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for flow cytometry and proteome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSTEMI: Patients presenting with a myocardial infarction will have blood samples taken for analysis. At the time of their angiography/angioplasty procedure they will have an OCT assessment of the culprit coronary artery to distinguish if the heart attack was caused by a plaque rupture or plaque erosion event
  Interventions: Diagnostic Test: Optical Coherence Tomography (OCT)
- Control: Patients undergoing planned angioplasty will have blood samples taken pre and post angioplasty to help as a control for the flow cytometry and for biomarker analysis

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography (OCT) — Optical Coherence Tomography (OCT) can undertake detailed characterisation of plaque morphology in patients with myocardial infarction at the time of percutaneous treatment. This allows plaque rupture, erosion and other mechanisms of myocardial infarction to be differentiated
  Groups: NSTEMI

SUMMARY:
Plaque erosion is associated with myocardial infarction (MI) in about 30% of cases and may require a different management approach to plaque rupture. The investigators hypothesise that plaque erosion leads to higher levels of apoptotic circulating endothelial cells (CECs) compared to plaque rupture.

Aims: To compare associations between plaque erosion and plaque rupture with numbers and types of apoptotic CECs in patients with non-ST elevation MI (NSTEMI) and stable coronary artery disease controls (CAD). Additional aims are to explore signals of cellular stress (mitochondrial dsDNA), sub-populations of activated neutrophils, circulating endothelial progenitor cells and erosion-specific plasma biomarkers.

Methods: Prospective observational study of 80 patients with NSTEMI and 40 patients with stable CAD. Plaque erosion or rupture will be identified by intracoronary Optical Coherence Tomography (OCT). CECs and neutrophils will be quantified and characterised using flow cytometry looking at markers of cell death and neutrophil activation. Plasma will be analysed by proteomic methods (Olink) and for mitochondrial dsDNA.

Potential importance of findings: This study will provide evidence for the hypothesised mechanism of plaque erosion and clarify if biomarker analysis in NSTEMI patients provides a basis for non-invasive diagnosis of plaque erosion versus rupture.

DETAILED DESCRIPTION:
This is a prospective observational pilot study to assess the feasibility of studying endothelial cell and neutrophil differences between coronary atherosclerotic plaque rupture and plaque erosion in patients presenting with NSTEMI. The data obtained from this study will be used to determine the feasibility of a larger study, if appropriate.

Patients presenting with a diagnosis of NSTEMI within 24 hours of chest pain will be approached to take part in the study if an invasive strategy is planned. A control group of patients scheduled to undergo elective PCI for stable angina will also be recruited.

Following written informed consent peripheral venous blood samples will be taken as soon as possible after admission (or immediately prior to elective PCI in the control group) this will be analysing using flow cytometry to determine circulating cell sub-populations. Stored plasma will be used for proteomic analysis (separate funding to be sought). Cellular populations will be isolated and characterised by transcriptome analysis using RNA-seq (separate funding to be sought).

The culprit lesion will be identified by coronary angiography in the NSTEMI group, and if feasible OCT will be undertaken in the culprit and non-culprit vessels. If OCT is not feasible (eg lesion requires pre-dilatation with a balloon, or vessel is too tortuous) the patient will be excluded from the study and no further study related procedures will be undertaken. Blood samples from such patients will also be discarded.

OCT data will be analysed off line by two independent experts to classify plaque morphology (rupture, erosion, other). Endothelial cell populations will be analysed in coronary and peripheral arterial blood using flow cytometry: results will be analysed according to OCT-defined plaque pathology.

Blood samples will be stored with a view to proteomic analysis using the Olink Cardiovascular panel.

The patients will be contacted at 1 month by telephone to determine vital status and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent, < 75 years old
* NSTEMI group: Admission to hospital within 24 hr of pain onset. Scheduled to undergo invasive angiography ± PCI during index admission
* Stable angina group: Scheduled to undergo elective PCI

Exclusion Criteria:

* Cardiogenic shock or haemodynamic instability,
* NSTEMI due to stent thrombosis restenosis, coronary dissection or embolism
* Previous CABG
* Requirement for mechanical ventilation
* Known severe renal impairment (eGFR <45 ml/min/1.73m2)
* Known haematological malignancy or systemic inflammatory disorder
* Requirement for emergency cardiac surgery
* Inability to carry out OCT

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All comers myocardial infractions/stable angina cases to the NNUH Cardiology team
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Apoptotic circulating endothelial cells | 1 year
  The hypothesis is that plaque rupture myocardial infarctions are correlated with higher levels of circulating endothelial cells (100-1000 cells per ml) in blood compared to levels seen following a plaque rupture myocardial infarction (less than 100 cells per ml).To measure these levels, plasma will be taken from patient and a sample analysed using flow cytometry to determine the levels of circulating endothelial cells. Invasive assessment of their coronary arteries at the time of angioplasty with an OCT scanner will differentiate the patients cause of heart attack into plaque eruption or plaque rupture.

SECONDARY OUTCOMES:
Neutrophils | 1 year
  It has been shown in models that TLR2 on neutrophils is required for the formation of an erosion-like coronary plaque. Using blood samples to quantify numbers of neutrophils via flow cytometry whilst also looking at which of these population are positive for TLR2 (TLR2 activation encourages further expression of TLR2). This is feasibility data to see whether human plaque erosion myocardial infarctions are associated with TLR2 positive neutrophils as in the models. Invasive assessment of their coronary arteries at the time of angioplasty with an OCT scanner will differentiate the patients cause of heart attack into plaque eruption or plaque rupture.
Endothelial progenitor cells | 1 year
  Endothelial Progenitor Cells (EPC) are a bone marrow derived cell line, the levels in blood at the time of a myocardial infarction correlate with a better prognosis from the myocardial infarction. Early EPCs (differentiated on flow cytometry CD34- / CD133+ / CD45+ / KDR+) have a paracrine function and promote angiogenesis. Late EPCs (differentiated on flow cytometry by CD34+ / CD133- / CD45dim / KDR+) can differentiate into endothelial cells. To measure the levels of EPCs (early and late) in blood of patients presenting with plaque erosion/rupture (as classified by OCT scanning at the time of angiography) and hypothesise plaque erosions will have higher levels (cells/ml) of these progenitor cells.
Biomarker analysis | 1 year
  At present it is only possible to differentiate plaque erosion from plaque rupture at a post-mortem examination or by invasive OCT assessment. Biomarker differences (using cytokine arrays) between patients with plaque rupture and plaque erosion myocardial infarctions have levels of TSP-1 and EGF in peripheral blood correlated with plaque rupture, whereas levels of I-TAC positively correlate with plaque erosion. Frozen plasma samples taken peripherally will have further array (OLink Cardiovascular panel 3) to see if any of these molecules correlate with plaque erosion/rupture. Further validation will be sought through ELISA assessments. Invasive assessment of their coronary arteries at the time of angioplasty with an OCT scanner will differentiate the patients cause of heart attack into plaque eruption or plaque rupture. OLink panels do not give a level of the molecule in blood only a differential of the differences in cytokine levels.

CONTACTS AND LOCATIONS:
Overall Officials: James Wardley, Principal Investigator — Specialist Trainee in Cardiology
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No